CLINICAL TRIAL: NCT00434668
Title: Randomized Phase II Study Evaluating The Tolerability Of Adjuvant Docetaxel-based Chemotherapy For Completely Resected Stage IB-II Non-Small Cell Lung Cancer (NSCLC): Toledo Trial
Brief Title: Evaluation of Tolerability of Adjuvant Cisplatin/Docetaxel in Completely Resected Stage IB/II Non-Small Cell Lung Cancer
Acronym: TOLEDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other); Sanofi (Industry)
Responsible Party: Prof Dr P Germonpré, Thoracale Oncologie Groep Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOGA 0501; Eudra CT 2005-004029-24
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Adjuvant chemotherapy for completely resected NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel; Vinorelbine

INTERVENTIONS:
Drug: cisplatin/docetaxel
Drug: cisplatin/vinorelbine

SUMMARY:
The aim of this study is to evaluate the tolerability (in terms of drug delivery and toxicity) of four cycles of adjuvant docetaxel plus cisplatin in patients with completely resected stage IB-II Non-Small Cell Lung Cancer. To avoid a selection bias, eligible patients will be randomised to receive cisplatin/docetaxel or cisplatin/vinorelbine.

ELIGIBILITY:
Inclusion Criteria:

* completely resected pathological stage IB or II NSCLC
* adequate haematological, renal and liver function and condition

Exclusion Criteria:

* previous chemo or radiotherapy for NSCLC
* bronchoalveolar cell subtype
* second active primary malignancy or serious concomitant medical disease
* difficulties with adequate follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2005-12; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Success of delivery treatment; data collected during chemotherapy treatment
Toxicity (occurrence of any grade 4 toxicity); data collected at the end of each cycle

SECONDARY OUTCOMES:
Overall toxicity
Progression free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Paul R. Germonpre, MD PhD, Principal Investigator — Universiteit Antwerpen
Locations (3):
- Belgium (3):
  - ZNA Middelheim, Antwerp, Antwerp
  - University Hospital Antwerp, Edegem, Antwerp
  - St Augustinus ziekenhuis, Wilrijk, Antwerp